CLINICAL TRIAL: NCT05119257
Title: (Bispecific) Antibodies in Cancer Patients (InHeAb01)
Brief Title: (Bispecific) Antibodies in Cancer Patients
Acronym: InHeAb01
Status: Available | Type: Expanded Access
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Helmut Salih, Head of CCU Translational Immunology (Developer and Manufacturer of applied bispecific antibodies), University Hospital Tuebingen
Other Study IDs: InHeAb01
Record Dates: First submitted 2021-10-18; First posted 2021-11-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Antibodies, Bispecific

STUDY DESIGN:
Expanded Access Types: Individual, Intermediate

INTERVENTIONS:
Biological: Bispecific antibodies (bsAB) — BsAbs equipped with a target-specificity directed to a TAA and an effector-specificity for an activating receptor on T cells, such as CD3 or CD28, are applied intravenously in repeated cycles until disease progression or dose limiting toxicity.

SUMMARY:
The aim of this project is to provide (bispecific) antibodies to individual patients with advanced solid and hematological malignancies without any available approved treatment options.

DETAILED DESCRIPTION:
Ethics: Patient treatment will be conducted according to §13 Absatz 2b, AMG (German law).

All (bispecific antibodies) applied are developed and manufactured by the principle investigator Prof. Helmut Salih.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of advanced malignant disease
* Advanced malignant disease without any available standard of care treatment option
* Live expectancy > 3 month
* Ability to understand and voluntarily sign an informed consent form.
* Ability to adhere to the visit schedule and other protocol requirements
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.

Exclusion Criteria:

* Pregnant or lactating females.
* Treatment regimens inducing severe T cell deficiencies
* Treatment-related side effect from prior cancer treatment > CTC grade 2 (CTCAE V5.0)
* Participation in any clinical study or having taken any investigational therapy, which would interfere with the studys primary and secondary end points within 2 weeks prior to Ab treatment.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- See also: CCU Translational Immunology — https://www.medizin.uni-tuebingen.de/de/das-klinikum/einrichtungen/kliniken/medizinische-klinik/kke-translationale-immunologie